CLINICAL TRIAL: NCT06297174
Title: A Single Dose, Randomized, Open-label, Two-treatment, Four-period, Two-sequence, Replicate Crossover Bioequivalence Study of Generic Racecadotril 100 mg Capsules and Reference Product (HIDRASEC®) in Healthy Thai Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Generic Racecadotril 100 mg Capsules Under Fasting Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharma Nueva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BE23-035
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Healthy Vollunteer
Keywords: Racecadotril; Bioequivalence study
MeSH Terms: interventions — racecadotril

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic Racecadotril 100 mg Capsules (Experimental): Generic Racecadotril 100 mg Capsules (test drug)
  Interventions: Drug: Racecadotril 100 mg Capsules; Drug: HIDRASEC®
- HIDRASEC® (Active Comparator): HIDRASEC® (Racecadotril 100 mg Capsules (reference drug))
  Interventions: Drug: Racecadotril 100 mg Capsules; Drug: HIDRASEC®

INTERVENTIONS:
Drug: Racecadotril 100 mg Capsules — Racecadotril 100 mg Capsules (test drug)
Drug: HIDRASEC® — HIDRASEC® (reference drug)
  Other Names: Racecadotril 100 mg Capsules

SUMMARY:
Objectives:

To determine and compare the rate and extent of absorption of a test formulation with that of a reference innovator formulation when given as equal labeled dose in healthy subjects under fasting conditions

Study Design:

An open label, randomized, two-treatment, four-period, two-sequence, replicate crossover bioequivalence study in healthy Thai volunteers under fasting conditions with at least 7 days washout period between the administrations of investigational products of each period

DETAILED DESCRIPTION:
Each subject will receive a single dose of racecadotril 100 mg capsules, as a test formulation (T) or a single dose of racecadotril 100 mg capsules, HIDRASEC, as a reference formulation (R), with 240±2 mL of ambient temperature drinking water after an overnight fasting for at least 10 hours. Investigational product will be provided to subject in stainless steel cup and subject will be dosed without touching the capsule. This activity will be followed by a mouth check using a tongue depressor and a flashlight to assess the compliance of dosing. The formulations will be given in a crossover fashion as per the randomization schedule. The dosing processes will be conducted under normal light condition.

In each period, total of 23 blood samples will be collected from 23 sampling time points. Blood samples (3.5 mL each) will be collected at time 0.00 (pre-dose) and at 0.16, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 24.00 and 36.00 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai male or female subjects between the ages of 18 to 55 years.
2. Body mass index between 18.5 to 30.0 kg/m2.
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.

   Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study.
4. Non-pregnant woman (negative pregnancy test) and not currently breast feeding.
5. Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 7 days after the end of study in Period 4. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:

   * Postmenopausal for at least 1 year or
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) at least 6 months
6. Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 4.
7. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria:

1. History of allergic reaction or hypersensitivity to the active substance or to any of the excipients.
2. History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hyper/hypothyroidism, diabetes mellitus), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hyper/hypotension), psychiatric (e.g. depression), neurologic (e.g. convulsion), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness.
3. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19.
4. History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
5. History or evidence of angioedema.
6. History of febrile illness within 7 days prior to check-in in each period.
7. History or evidence of antibiotic-associated colitis such as pseudomembranous colitis.
8. History or evidence of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
9. History of problems with swallowing tablet or capsule.
10. History of sensitivity to heparin or heparin-induced thrombocytopenia.
11. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy.
12. History of diarrhea, dehydration or vomiting within 24 hours prior to check-in in each period.
13. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine).
14. Investigation with blood sample shows positive test for HBsAg.
15. Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test.
16. History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study.
17. History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.).
18. History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result.

    In case of alcohol breath test result represents the alcohol concentration range of 1 - 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC.
19. History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study.
20. Consume or drink juice of grapefruit or orange or pomelo or its supplement/containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study.
21. Use of prescription or nonprescription drugs (e.g. paracetamol, ACE inhibitors, other drug that can induced angioedema such as angiotensin II receptor blockers, direct renin inhibitors, betalactam antibiotics and other non-steroidal anti-inflammatory drugs (NSAIDs), etc.), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study.
22. Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study.
23. Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment.
24. Subjects with poor venous access or intolerant to venipuncture.
25. Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study.
26. Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team.
27. Subjects who are employees of International Bio Service Co., Ltd., Pharma Nueva Co., Ltd. or Siam Pharmaceutical Co., Ltd.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2024-09-17 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Plasma area Under the Curve (AUC(0-36hr)) for Racecadotril | Through 36 hours post dose
  Plasma area Under the Curve (AUC(0-36hr)) for Racecadotril
Peak Plasma Concentration (Cmax) of Racecadotril | 36 hours post dose
  Peak Plasma Concentration (Cmax) of Racecadotril

CONTACTS AND LOCATIONS:
Overall Officials: Porranee Puranajoti, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No
Confidential